CLINICAL TRIAL: NCT05440175
Title: Effects of Combined Electrical Muscle Simulator and Mirror Therapy in Upper Limb Stroke Patients
Brief Title: Effects of Combine EMS and Mirror Therapy in Upper Limb Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nouman Khan (Other)
Responsible Party: Sponsor-Investigator, Nouman Khan, lecturer, Shifa Tameer-e-Millat University
Organization: Shifa Tameer-e-Millat University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sabahat IRB #351-21
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Stroke
Keywords: Electrical muscle stimulation; Constraint induced movement therapy; Mirror therapy
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy; Exercise

STUDY DESIGN:
Intervention Model Description: This is an randomized control trail in which the stroke patients are divided into three different treatment group.
Who Masked: Participant
Masking Description: The participant were blinded about the treatment group in which they are enrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): The participants will be given Mirror therapy along with the electrical muscle stimulation and exercises.
  Interventions: Other: EMS, Mirror therapy & exercises
- Group B (Experimental): The participants will be given constraint induced movement therapy (CIMT) along with exercises.
  Interventions: Other: CIMT & exercises
- Group C (Experimental): The participants will be given mirror therapy and exercises.
  Interventions: Other: Mirror therapy & exercises

INTERVENTIONS:
Other: EMS, Mirror therapy & exercises — EMS will be applied with frequency between 20-100 Hz and pulse width between 20 to 450us and Mirror therapy for 30 minutes and four days per week for a total duration of 12 weeks. Exercises include the flexion, extension of the wrist and elbow, ulnar and radial deviations , place any cylindrical object in patients palm and ask to lift the object off the table. other exercises includes external and internal rotations with different task orientations.
  Arms: Group A
Other: CIMT & exercises — Constraint induced movement therapy will be applied for 30 minutes and four days per week for a total duration of 12 weeks, it is a form of rehabilitation therapy that improves upper limb movement, it claims to improve the arm motor ability and the functional use of a paretic arm- hand. Exercises include the flexion, extension of the wrist and elbow, ulnar and radial deviations , place any cylindrical object in patients palm and ask to lift the object off the table. other exercises includes external and internal rotations with different task orientations.
  Arms: Group B
Other: Mirror therapy & exercises — Mirror therapy will be given for 30 minutes and four days per week for a total duration of 12 weeks. The exercises include the flexion, extension of the wrist and elbow, ulnar and radial deviations , place any cylindrical object in patients palm and ask to lift the object off the table. other exercises includes external and internal rotations with different task orientations.
  Arms: Group C

SUMMARY:
This study will be designed to evaluate the effectiveness mirror therapy combined with electrical muscle stimulations compared with constraint induced therapy in upper limb stroke patients. The aim of the study is to investigate the therapeutic effectiveness of mirror therapy and EMS in stroke patients and compare the outcomes with CIMT.

DETAILED DESCRIPTION:
Stroke or CVA is the sudden death of the brain cells due to inadequate blood flow, it's a focal disturbance of cerebral function, with symptoms lasting for 24hrs or longer or leading to death, with no apparent cause other than of vascular origin. The commonest consequence of stroke is loss of upper limb function. The protocol planned for improving the function of the upper limb is mirror therapy combined with EMS and compare with constraint-induced movement therapy (CIMT) treatment in stroke patients Many works done on CIMT and mirror therapy in rehabilitation prove to be powerful tools for upper limbs in people with stroke. Different studies concluded that CIMT is more effective than Mirror Therapy (MT) in the upper extremity in stroke patients. An RCT was published in 2019 in which mirror therapy combined with electrical stimulation proves to be effective in stroke patients. However, I have not found a study comparing EMS combined with Mirror therapy compared to CIMT treatment in stroke patients. According to the Alternate hypothesis mirror therapy combined with EMS has beneficial effects on clinical outcomes in upper limb stroke patients. According to the null hypothesis, CIMT has better results in stroke patients as compared to EMS combined with Mirror therapy.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female stroke patients above 45 years
* Ischemic and Haemorrhagic chronic stroke patients
* Participants should be able to do 100 wrist extension

Exclusion Criteria:

* Patients with an implanted electrical device
* Patients with paresis
* Patients of hemiplegia caused due to other brain injuries (TBI, tumour), Coordination problem
* Individuals with impaired sensory perception

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Fugl- Meyer Assessment | 12 weeks
  Fugl- Meyer Assessment scale is a stroke specific performance- based impairment index. it has 226 total score and has 5 domains to assess the motor functions, overall reliability of FMA scale was high overall intraclass correlation coefficient varies from 0.61 to 0.97 for the upper extremity and the validity coefficient ranged from 0.91 to 0.97.

SECONDARY OUTCOMES:
Motor assessment scale | 12 weeks
  motor assessment scale is a stroke-specific scale that includes 7 points from 0-6 which includes tone and optimal behavior. A score of 4 on this item indicates a consistently normal response, a score > 4 indicates persistent hypertonus, and a score < 4 indicates various degrees of hypotonus.

CONTACTS AND LOCATIONS:
Overall Officials: sabahat zahid chaudhary, DPT, Principal Investigator — Students
Locations (1):
- Shifa tameer e millat university, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee D, Lee G. Effect of afferent electrical stimulation with mirror therapy on motor function, balance, and gait in chronic stroke survivors: a randomized controlled trial. Eur J Phys Rehabil Med. 2019 Aug;55(4):442-449. doi: 10.23736/S1973-9087.19.05334-6. Epub 2019 Mar 22. PMID 30916531